CLINICAL TRIAL: NCT00756288
Title: A Randomized Controlled Paired Comparison of Photo-therapy With a Topical Retinoid Cream Pretreatment Versus PDT Alone for Actinic Keratoses
Brief Title: Photo-therapy With a Topical Retinoid Versus Photo-therapy Alone for Actinic Keratoses
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Associate Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU2574
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Actinic Keratoses
Keywords: Actinic Keratoses; Blue light therapy; photosensitizer; Retinoid
MeSH Terms: conditions — Keratosis, Actinic | interventions — Retinoids; Phototherapy; Photosensitizing Agents; Photochemotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Topical retinoid and Light therapy with photosensitizing agent
  Interventions: Procedure: Topical retinoid and blue-light therapy with photosensitizing agent
- 2 (Active Comparator): Light therapy with photosensitizing agent
  Interventions: Procedure: Photodynamic Therapy (PDT)

INTERVENTIONS:
Procedure: Topical retinoid and blue-light therapy with photosensitizing agent — Topical Retinoid - Apply to AKs for 4 weeks Photo-therapy with photosensitizing agent- Apply to AKs at week 4
  Arms: 1
Procedure: Photodynamic Therapy (PDT) — Photo-therapy with sensitizing agent - apply to AKs at week 4
  Arms: 2

SUMMARY:
Evaluating safety and efficacy of the use of topical retinoid with photodynamic therapy for the treatment of actinic keratoses.

DETAILED DESCRIPTION:
Evaluating safety and efficacy of the use of topical retinoid with photodynamic therapy vs photodynamic therapy alone for the treatment of actinic keratoses.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18-80 years old
* Subjects with AK lesions who will receive PDT
* Subjects with AK lesions in two areas other than face and scalp each with a surface area of 10cm2 or greater and at least 3 clinically diagnosed non-hypertrophic AK lesions in each
* Subjects in good health
* Subjects with willingness and the ability to understand and provide informed consent

Exclusion Criteria

* Subjects who are pregnant or lactating
* Subjects with a history of cutaneous photosensitivity or porphyria, hypersensitivity to porphyrins, or photodermatosis
* Subjects with use of photosensitizing drugs within 1 week of study start
* Subjects with use of topical medications such as corticosteroids, alpha-hydroxyacids or retinoids 2 weeks before study entry
* Subjects who received previous treatment of target AKs within 4 weeks
* Subjects who are unable to understand the protocol or give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Live blinded rater and blinded photo rater analysis of areas at week 0 and week 6 for erythema, edema, crusting, ulceration, palpability, need to cease/delay treatment, and overall response in reduction of number of actinic keratoses (AKs). | 6 weeks

SECONDARY OUTCOMES:
Subjects will assess pain, burning and itching on a scale of 0-3 at week 0, during retinoid treatment, during photo-therapy, one day after, and week 6. Also, principal investigator will evaluate adverse events at week 6. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University Department of Dermatology